CLINICAL TRIAL: NCT03898570
Title: Distributed Registry Study
Brief Title: Distributed Registry
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB-47517
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication; Arteriosclerosis; Atherosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases; Peripheral Vascular Diseases; Signs and Symptoms; Patient Compliance
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Arteriosclerosis; Atherosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases; Peripheral Vascular Diseases; Signs and Symptoms; Patient Compliance | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing vascular surgery procedures: Patients will report outcomes via their smartphone.
  Interventions: Behavioral: Patient reported outcomes

INTERVENTIONS:
Behavioral: Patient reported outcomes — Patients will download the research app onto their phone and enter pertinent medical history and surgical history data similar to standard registries for specific procedures. Over the next 12 months the investigators will obtain patient-reported outcomes (PROs) using the patient's phone.
  Specifically, the investigators will obtain daily activity data, weekly 6-minute-walk tests, and quarterly quality of life surveys

SUMMARY:
The purpose of this study is to test if a patient can be directly connected to a quality assurance (QA) database, traditionally known as a registry. Patient-reported outcomes (PRO) data will be entered into the database directly from a patient's mobile phone from their index procedure for 12 months. The investigators hope this study to be a "proof of concept" for such a distributed registry and evaluate 1) consistency of data acquisition, 2) engagement of patients, 3) overall value of patient-reported outcomes to enhance long term follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cardiovascular disease who are scheduled or have undergone either a) open or endovascular vascular procedure, or b) open or percutaneous cardiac procedure.
2. Patients with smartphones (iOS or Android) with unlimited data plans.
3. Patients who agree to remote surveillance

Exclusion Criteria:

1. Patients unwilling to download a research study app.
2. Data plans which are not unlimited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults with an iPhone 5s or higher who can read English
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcomes (PROs) using mobile app | 1 Year
  PROs are any report of the status of a patient's health condition that comes directly from the patient, without interpretation of the patient's response by a clinician or anyone else

CONTACTS AND LOCATIONS:
Overall Officials: Oliver O Aalami, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Palo Alto Veterans Hospital, Palo Alto, California
  - Stanford, Palo Alto, California

IPD SHARING:
Plan to Share IPD: No